CLINICAL TRIAL: NCT04223713
Title: Changes of Aortic Flow Patterns Detected by 4D- Flow- MRI After Trileaflet Reconstruction of the Aortic Valve With Autologous Pericardium Compared to Prosthetic Valve Replacement With Biological Prosthesis
Brief Title: 4D- Flow- MRI After Aortic Valve Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 77/19-S
Record Dates: First submitted 2019-11-29; First posted 2020-01-10 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-01

CONDITIONS: Aortic Valve Disease
Keywords: aortic stenosis; aortic regurgitation; Trileaflet reconstruction of the aortic valve; Biological aortic valve prosthesis; aortic flow patterns; MRI
MeSH Terms: conditions — Aortic Valve Disease; Aortic Valve Stenosis; Aortic Valve Insufficiency | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TriRec (Experimental): Trileaflet Reconstruction of the Aortic Valve
  Interventions: Procedure: TriRec
- Aortic valve replacement (Experimental): Biological prosthesis, Device: Edwards Perimount
  Interventions: Procedure: Aortic valve replacement

INTERVENTIONS:
Procedure: TriRec — Trileaflet Reconstruction of the Aortic Valve
  Arms: TriRec
Procedure: Aortic valve replacement — Biological Prosthesis, Device: Edwards Perimount
  Arms: Aortic valve replacement

SUMMARY:
This randomized controlled trial was designed to analyze flow patterns in the ascending aorta with MRI after either Trileaflet reconstruction of the aortic valve with autologous pericardium (TriRec) or surgical valve replacement with biological prosthesis. The hypothesis is that after TriRec procedure more physiological flow patterns will be observed, compared to biological valve prosthesis.

DETAILED DESCRIPTION:
Trileaflet reconstruction of the aortic valve with autologous pericardium (TriRec) is a new treatment option for diseased aortic valves and offers benefits compared to conventional valve replacement. At the moment no prospective randomized trials evaluating the role of the TriRec procedure are available and factors contributing to long- term durability are unknown.

The investigators want to examine aortic flow patterns with 4D- Flow- Magnetic Resonance Imaging (MRI) in patients after the TriRec procedure or biological prosthetic valve replacement in a prospective randomized trial. Flow patterns in the ascending aorta, examined with 4D- Flow- MRI, show nearly laminar flow patterns and no outflow obstruction in healthy subjects with tricuspid aortic valves. In contrast, helical flow patterns, turbulences and increased flow velocities are observed in diseased valves and also after valve replacement with mechanical or biological prostheses. These helical flow patterns seem to influence aortic wall remodeling and may contribute to structural valve dysfunction of biological prosthesis.

The investigators hypothesize that after TriRec procedure more physiological flow patterns will be observed, compared to biological valve prosthesis. The results can contribute to understand mechanisms for long- term performance of this technique and determine the role of this novel technique for treatment of aortic valve disease.

ELIGIBILITY:
Inclusion Criteria:

* Age > 50 years
* Documented symptomatic moderate or greater aortic stenosis or severe aortic insufficiency
* Aortic annulus > 19 mm
* Written informed consent of the patients.

Exclusion Criteria:

* Concomitant intervention of the aortic root, ascending aorta or aortic arch
* Concomitant valve surgery
* Emergency surgery for any reason
* Neurological events (i.e. stroke, TIA) within the previous 6 months
* Coagulation disorders (including thrombocytopenia < 100.000/ml)
* Porcelain aorta/severe calcification of the ascending aorta
* Active endocarditis or other active systemic infections
* Participating in another trial that may influence the outcome of this trial
* Pregnancy
* Dual antiplatelet therapy
* Previous cardiac surgery (excluding percutaneous procedures)
* Contraindication for MRI- examinations

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-01-14 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Flow velocity in the ascending aorta (m/s) | Day 4-7 post surgery
  Flow velocity in meters/ second in the ascending aorta in patients receiving either TriRec or biological prosthetic valve replacement measured by 4D- Flow- MRI.

SECONDARY OUTCOMES:
Flow vortices | Day 4-7 post surgery
  Flow vortices: defined as rotating particles around a point within the vessel with the rotational direction diverting > 90° from the physiological flow direction.
Flow helicality | Day 4-7 post surgery
  Blood revolving around an axis parallel to the main blood flow generating a corkscrew like figure
Systolic eccentricity | Day 4-7 post surgery
  Localization of the main blood flow vector (central, little, severe eccentricity).
Flow patterns in the left ventricular outflow tract. | Day 4-7 post surgery
  Flow patterns in the left ventricular outflow tract.
Effective orifice area (4D-Flow-MRI) | Day 4-7 post surgery
  Effective orifice area (cm2) of the reconstructed or replaced valve (4D- Flow- MRI)
Effective orifice area (TTE) | Day 4-7 post surgery
  Effective orifice area (cm2) of the reconstructed or replaced valve (transthoracic echocardiography (TTE)
Peak- and mean pressure gradients (mmHg, TTE) | Day 4-7 post surgery
  Peak- and mean pressure gradients (mmHg, TTE)
Left- ventricular diameters (mm, TTE) | Day 4-7 post surgery
  Left- ventricular diameters (mm, TTE)
Left- ventricular ejection fraction (%, TTE) | Day 4-7 post surgery
  Left- ventricular ejection fraction (%, TTE)
Quantification of aortic regurgitation (MRI) | Day 4-7 post surgery
  Quantification of aortic regurgitation (MRI)
Quantification of aortic regurgitation (TTE) | Day 4-7 post surgery
  Quantification of aortic regurgitation (TTE)

CONTACTS AND LOCATIONS:
Locations (1):
- Deutsches Herzzentrum Muenchen, Department of Cardiovascular Surgery, Munich, Germany